CLINICAL TRIAL: NCT01442454
Title: Endoscopic Ultrasound (EUS) Features of Chronic Pancreatitis: A Prospective Correlation With Intraoperative Findings and Surgical Pathology
Brief Title: Endoscopic Ultrasound (EUS) Features of Chronic Pancreatitis
Status: Terminated | Type: Observational
Why Stopped: The PI left and then the PI who would be taking over has left. No other investigator wanted to take the study since not sponsored
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 1008-15
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Pancreatitis
Keywords: chronic pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Pancreatitis
  Interventions: Other: chronic pancreatitis

INTERVENTIONS:
Other: chronic pancreatitis — No intervention, subjects followed through surgery

SUMMARY:
The purpose of this study is to correlate Endoscopic Ultrasound (EUS) criteria for chronic pancreatitis with surgical pathology.

ELIGIBILITY:
Patients who are eligible are individuals who have:

* normal pancreas
* suspected chronic pancreatitis
* established chronic pancreatitis (by ERCP, MRI, previous EUS, CT)
* pancreatic cancer

Patients who are not eligible are individuals who have:

• an uncorrectable coagulopathy (platelet <50,000, INR>1.5), or bleeding disorder, or are unable to discontinue anticoagulation 5-7 days prior to EUS (aspirin and bridging therapy with lovenox are allowed, clopidogrel is not allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing EUS
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States